CLINICAL TRIAL: NCT01125254
Title: Amlodipine Use in the Prevention and Treatment of Iron Overload in Patients With Thalassemia Major
Acronym: AnloThal
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Juliano de Lara Fernandes, Research Physician, University of Campinas, Brazil
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 000002
Record Dates: First submitted 2010-05-13; First posted 2010-05-18 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2015-01

CONDITIONS: Thalassemia Major
Keywords: thalassemia major; calcium channel blockade; magnetic resonance imaging
MeSH Terms: conditions — beta-Thalassemia | interventions — Amlodipine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amlodipine (Experimental): amlodipine 5mg qd
  Interventions: Drug: Amlodipine
- Controls (Placebo Comparator): placebo
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Amlodipine — 5mg po for 12 months

SUMMARY:
This study aims to investigate the use of amlodipine, a drug that blocks the uptake of calcium into cells, in the prevention and treatment of iron overload in patients with thalassemia major. Since iron uses the same calcium channels to enter the heart, pancreas and other organs, blocking these channels might help to prevent the accumulation of iron in these tissues. The study will follow 10 patients with thalassemia major: 5 will openly receive amlodipine and 5 will serve as controls, not receiving any additional drugs. Patients will be monitored through one year with an additional year of follow up after the group using amlodipine stops its use. Monitoring will occur through the measurement of blood ferritin as well as live and heart T2* by MRI.

ELIGIBILITY:
Inclusion Criteria:

* patients with thalassemia major over 6 years of age in use of iron chelating therapy.

Exclusion Criteria:

* pregnancy;
* advanced heart failure with NYHA III/IV or LVEF < 35%;
* formal contra-indications to an MRI study;
* patient with advanced heart block.

Ages: 6 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Myocardium T2* | 12 months
  Heart T2* by MRI at 12 months

SECONDARY OUTCOMES:
Liver T2* | 24 months
  Liver T2* by MRI every 6 months for 2 years. First year with active treatment; second year with withdrawal.
Heart volumes | 24 months
  Diastolic and systolic volumes by MRI every 6 months for 2 years. First year with active treatment; second year with withdrawal.
Left ventricle ejection fraction | 24 months
  LVEF by MRI every 6 months for 2 years. First year with active treatment; second year with withdrawal.
Serum ferritin | 24 months
  Serum ferritin every 6 months for 2 years. First year with active treatment; second year with withdrawal.
Myocardium T2* | 6-18-24 months
  Heart T2* by MRI every 6 months until 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Juliano L Fernandes, MD, Principal Investigator — University of Campinas, Brazil
Locations (1):
- University of Campinas, Campinas, São Paulo, Brazil

REFERENCES:
- [Derived] Padhani ZA, Gangwani MK, Sadaf A, Hasan B, Colan S, Alvi N, Das JK. Calcium channel blockers for preventing cardiomyopathy due to iron overload in people with transfusion-dependent beta thalassaemia. Cochrane Database Syst Rev. 2023 Nov 17;11(11):CD011626. doi: 10.1002/14651858.CD011626.pub3. PMID 37975597